CLINICAL TRIAL: NCT01700101
Title: MelaFind Evaluations for Patients With Multiple Nevi
Status: Completed | Type: Observational
Sponsor: MELA Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20123
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Clinically Atypical Pigmented Skin Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We have added objectives 4-6 to our updated study:

Study Objective 1: To determine whether the distribution of MelaFind scores is different for different patients with multiple nevi, and whether such distributions can be utilized to identify "signature" lesions for a given patient.

Study Objective 2: To investigate whether distributions of quantitative ABCD parameters differ among patients and whether these qABCD parameters identify "signature" lesions.

Study Objective 3: To determine the feasibility of defining and using relative thresholds to improve the specificity of MelaFind without sacrificing its high sensitivity.

Study Objective 4: To determine the repeatability of MelaFind scores for a given lesion for different patient and lesion characteristics.

Study Objective 5: To identify patient and lesion characteristics that result in the highest variability of MelaFind scores for a given lesion.

Study Objective 6: To use standard errors of MelaFind scores to propose a robust individual threshold for lesions to be considered for biopsy to rule out melanoma on patients with multiple nevi.

ELIGIBILITY:
Cutaneous lesions examined with MelaFind must satisfy all of the following inclusion criteria:

Inclusion Criteria:

* The lesion is pigmented (i.e., melanin, keratin, blood)
* The diameter of the pigmented area is not < 2 mm, and not > 22 mm
* The lesion is accessible to the MelaFind
* The patient, or a legally authorized representative, has consented to participate in the study and has signed the Informed Consent Form;

Cutaneous lesions that meet any of the following exclusion criteria will not be accepted:

Exclusion Criteria:

* The patient has a known allergy to isopropyl alcohol
* The lesion has been previously biopsied, excised, or traumatized
* The skin is not intact (e.g., open sores, ulcers, bleeding)
* The lesion is within 1 cm of the eye
* The lesion is on mucosal surfaces (e.g., lips, genitals)
* The lesion is on palmar hands
* The lesion is on plantar feet
* The lesion is on or under nails
* The lesion is located on or in an area of visible scarring
* The lesion contains foreign matter (e.g., tattoo, splinter, marker)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have at least one lesion that meets the inclusion/exclusion criteria (see eligibility criteria below) AND each lesion enrolled must be clinically atypical (i.e., contain at least one of the following ABCDEPRU characteristics: Asymmetry, Border irregularity, Color variegation, Diameter < 6 mm, Evolving, Patient's concern, Regression, Ugly duckling).
  Lesions should be selected to have characteristics that may affect the repeatability of lesion scores: anatomic site (often exposed to UV - sun or tanning beds - or not; sun-damage may affect the repeatability); lesion diameter (6 mm, e.g. ~5 mm or > 6 mm, e.g., 10 mm); and melanin content relative to normal skin (dark pigmentation or light pigmentation).
  A maximum of 8 lesions may be enrolled per patient
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Multiple values and standard deviations of MelaFind scores for pigmented skin lesions | 1 month